CLINICAL TRIAL: NCT00586521
Title: A Prospective Controlled Study on the Effect on Bleeding Events and Joint Function in Young Adults With Severe Hemophilia A After a 6 Month Prophylaxis Treatment Compared to on Demand Treatment
Brief Title: BAY14-2222 Prophylaxis and Joint Function Improvement (Adults)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11859; 2005-002757-45 (EudraCT Number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Hematologic Disease; Hemophilia A
Keywords: Coagulation Disorders
MeSH Terms: conditions — Hematologic Diseases; Hemophilia A; Hemostatic Disorders | interventions — F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rFVIII-FS (octocog-alfa), (Kogenate FS) (Experimental): On-demand treatment was to follow the same treatment pattern the subject was using before entering the study. While on prophylactic treatment, all subjects were to be treated at a dose of 20-40 IU/kg, 3 times per week at a stable dose.
  Interventions: Drug: Kogenate (BAY14-2222)

INTERVENTIONS:
Drug: Kogenate (BAY14-2222) — One group two treatment schedules, first on-demand then switch to prophylaxis

SUMMARY:
The purpose of the study is to evaluate the effect of prophylactic treatment on the number of joint bleeds and quality of life in severe hemophilia A subjects compared to on-demand treatment in a one-group two-treatment schedule design.

In addition, the effect of prophylactic treatment on the joint function, the number of all bleeds, and on the quality of life compared to on-demand treatment and health-economic data will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (< 1% FVIII)
* 30-45 years of age
* Previously treated subject (> 100 Exposure days to any FVIII)
* On-demand therapy with any FVIII

Exclusion Criteria:

* No history of inhibitor
* No planned elective orthopedic surgery during the study duration (13 months)
* No severe concomitant disease
* No history of anaphylactic or other severe reaction to previous FVIII treatment

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- United States (3):
  - Aurora, Colorado
  - Chapel Hill, North Carolina
  - Houston, Texas
- Strasbourg, France
- Italy (3):
  - Florence
  - Pavia
  - Roma
- Spain (2):
  - Madrid, Madrid
  - Santa Cruz de Tenerife, Santa Cruz de Tenerife
- United Kingdom (2):
  - Cardiff, South Glamorgan
  - Sheffield, South Yorkshire

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at Haemophilia treatment centers
Pre-assignment Details: All subjects who met eligibility criteria on screening were enrolled into the study and began the on-demand treatment period.
Period: On Demand Treatment (Months 1-6)
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Prophylactic Treatment (Months 8-13)
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Target joints presence [Number; unit: participants] — 16 (80%) subjects had at least 1 target joint; in most elbow(s) and/or ankles(s) were affected
  participants
    Number participants with target joints presence | 16
    Number participants without target joints presence | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Joint Bleeds
Description: Number of joint bleeds during Months 8-13 compared to number of joint bleeds during Months 1-6
Time Frame: Months 1-6 (on-demand treatment) and 8-13 (prophylactic treatment)
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: Number of joint bleeds
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Number analyzed (Participants) | 20
Number of joint bleeds
  Months 1-6 (on-demand) | 18.5 (11.6)
  Months 8-13 (prophylactic) | 1.5 (2.1)
Statistical Analysis 1: Comparison: rFVIII-FS (Octocog-alfa), (Kogenate FS); The primary outcome measure was analyzed by paired t-test and Wilcoxon test (number of joint bleeds prophylaxis treatment compared to number of joint bleeds on-demand treatment) at 6 months of treatment; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: rFVIII-FS (Octocog-alfa), (Kogenate FS); The maximum individual reduction in the actual number of joint bleeds after the switch to prophylactic treatment was analyzed by a paired t-test of the individual difference between prophylaxis treatment bleed compared to on-demand treatment bleeds; Test type: Superiority or Other; p < 0.001, paired t-test

2. Secondary Outcome: Number of All Bleeds
Description: Mean number of all bleeds during Months 8-13 (prophylactic) compared to mean number of all bleeds during Months 1-6 (on-demand)
Time Frame: Months 1-6 (on-demand treatment) and 8-13 (prophylactic treatment)
Population: intention-to-treat
Measure: Mean (Standard Deviation); unit: All bleeds
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Number analyzed (Participants) | 20
All bleeds
  Months 1-6 (on-demand) | 23.7 (13.3)
  Month 8-13 (prophylactic) | 1.9 (3.3)
Statistical Analysis 1: Comparison: rFVIII-FS (Octocog-alfa), (Kogenate FS); paired t-test (prophylaxis compared to on-demand) at 6 months of treatment; Test type: Superiority or Other; p < 0.001, paired t-test

3. Secondary Outcome: Physical Assessment Compared to On-demand Treatment as Determined by the Gilbert Score
Description: Total score with a range of 0-100, evaluating ankle, knee and elbow, 0 indicates normal function, higher values indicate joint damage
Time Frame: Month 13 (end of prophylactic treatment) and Month 6 (end of on-demand treatment)
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: Gilbert score (0-100)
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Number analyzed (Participants) | 20
Gilbert score (0-100)
  Month 6 (on-demand) | 25.3 (11.7)
  Month 13 (prophylactic) | 19.8 (11.7)
Statistical Analysis 1: Comparison: rFVIII-FS (Octocog-alfa), (Kogenate FS); The Gilbert Score was the sum of 3 scores: pain (0=no pain to 3=severe pain); bleeding score (0=none to 3=3 or more major bleeds or 7 or more minor bleeds); and physical score (based on swelling, muscle atrophy; and axial deformity (at knee or ankle), range of motion, crepitus on motion, flexion contracture, instability; Test type: Superiority or Other; p < 0.001, paired t-test

4. Secondary Outcome: Quality of Life Compared to On-demand Treatment as Measured by the Haemo-QoL A Questionnaire
Description: Total transformed score with a range of 0-100, higher values indicate better outcome. 41 items in 6 domains: physical functioning; role functioning; worry; consequences; positive affect; treatment concern.
Time Frame: Month 13 (end of prophylactic treatment) and Month 6 (end of on-demand treatment)
Population: intent-to-treat-population
Measure: Mean (Standard Deviation); unit: Transformed score
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Number analyzed (Participants) | 20
Transformed score
  Month 6 (on-demand) | 73.4 (17.4)
  Month 13 (prophylactic) | 75.9 (16.1)
Statistical Analysis 1: Comparison: rFVIII-FS (Octocog-alfa), (Kogenate FS); The Haemo-QoL A questionnaire measures the subject's self-assessment of disease impact on "physical functioning", "role functioning", "worry", "consequences", "positive affect", and "treatment concern"; Test type: Superiority or Other; p = 0.314, paired t-test — The alpha level for a significant P-value was pre-defined at 5%

ADVERSE EVENTS:
Arm/Group | rFVIII-FS (Octocog-alfa), (Kogenate FS)
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIII-FS (Octocog-alfa), (Kogenate FS) (N=20)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Alcohol use (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIII-FS (Octocog-alfa), (Kogenate FS) (N=20)
Lower respiratory tract infection (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Anxiety (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
The short observation period of 6 months may be responsible for the lack of statistical significance between treatments in the subject's overall assessment of disease-related quality of life; however, a positive trend was noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less